CLINICAL TRIAL: NCT04748978
Title: Office Preparation of Partially Intramural Uterine Myomas (OPPIuM) and Myolysis With Diode Laser Dual Wavelengths Laser System (DWLS) for the Treatment of G1-G2 Symptomatic Myomas
Brief Title: OPPIuM Technique and Myolysis With Diode Laser Dwls
Acronym: Myolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cagliari (Other)
Collaborators: University of Foggia (Other); Azienda Ospedaliera Ordine Mauriziano di Torino (Other); Civic Hospital, Italy (Other); Clinical Hospital Center Rijeka (Other); BelMedic Hospital, Beograd, Serbia (Unknown)
Responsible Party: Principal Investigator, Stefano Angioni, Full Professor, University of Cagliari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPPIuM MYOLYSIS DWLS
Record Dates: First submitted 2021-01-30; First posted 2021-02-10 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Uterine Fibroid; Myoma;Uterus
Keywords: fibroid; myoma; hysteroscopy; diode laser
MeSH Terms: conditions — Leiomyoma; Myofibroma; Myoma | interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- symptomatic uterine fibroids (Experimental): patients aged between 18 and 48 years with clinical and/or ultrasound diagnosis of uterine fibromatosis
  Interventions: Procedure: hysteroscopy

INTERVENTIONS:
Procedure: hysteroscopy — OPPIum and Myolysis
  Other Names: myolysis

SUMMARY:
PURPOSE OF THE STUDY The study aims to examine the feasibility and effectiveness of the OPPIuM technique combined with myolysis using the DWLS diode laser. In addition, to evaluate the reduction of myoma volume and the extent of uterine bleeding with myolysis to improve women's quality of life and avoid resectoscope hysteroscopy for a G2 MIOMA, which may lead to an increase in intraoperative surgical risks and long-term complications.

POPULATION 35 patients aged between 18 and 48 years with clinical and/or ultrasound diagnosis of uterine fibromatosis, belonging to the Endometriosis/Pelvic Chronic Pain Centre of the Complex Operating Unit of Gynecology of the University Polyclinic of Monserrato and other centers involved in the study. To be eligible for inclusion, patients with ultrasound and hysteroscopic diagnosis of a single submucosal myoma, partially intramural (G1 or G2) ≤ 3 cm, must present symptoms such as abnormal uterine bleeding and pelvic pain, for which surgical treatment was scheduled.

INCLUSION CRITERIA

* Women between 18 and 48 years old
* Diagnosis of symptomatic uterine fibromatosis (abnormal uterine bleeding and/or pelvic pain) with single fibroma ≤ 3 cm G1 or G2.

EXCLUSION CRITERIA Patients who cannot provide written informed consent or follow the procedures set out in the protocol.

* Patients with malignant neoplasms or serious systemic diseases
* Patients with multiple fibroids or single > 3 cm
* Asymptomatic patients
* Patients with other uterine or related diseases
* Patients seeking a pregnancy. INTERVENTION STRATEGY AND INSTRUMENTS

A total of 35 women will initially be included in the study, of which:

Patients will undergo the following assessments:

* Collection of physiological, pathological, and pharmacological anamnesis
* Collection of diagnostic tests (ultrasound) and staging of the underlying disease (uterine fibromatosis)
* Completion of the PBAC questionnaire
* Transvaginal ultrasound
* Office diagnostic hysteroscopy with OPPIuM and Myolysis
* Possible resectoscope hysteroscopy or laser myomectomy in narcosis.

DETAILED DESCRIPTION:
BACKGROUND Leiomyomas or uterine fibroids are benign lesions that can cause infertility, uterine bleeding (hypermenorrhea, metrorrhagia, and menometrorrhagia), resulting in anemia, disorders in urinary tract function and symptoms of abdominal pressure, chronic pelvic pain, and/or dysmenorrhea. Often doctors decide to remove the myoma or uterus to resolve the symptoms. Myomas or uterine fibroids occur in 25 to 44% of women during reproductive age. Myomas are more common in the fourth and fifth decade of life when their incidence can reach almost 70% in Caucasian women and over 80% in African origin women.

Submucosal fibroids are classified according to their development within the endometrial cavity in G0: intracavitary pedunculate fibroids G1 : fibromas whose intramural development is less than 50%. G2 : fibromas whose intramural development is greater than or equal to 50%. Resectoscope myomectomy for G2 myomas is a difficult procedure that should only be performed by surgeons experienced in hysteroscopy. In fact, resectoscope hysteroscopy is associated with a significant risk of complications that is proportional to the degree of intramural development of the myoma. Furthermore, the greater the myoma and its intramural development, the more likely the procedure will need to be divided into several surgical interventions.

As a result of these problems, several myolysis techniques have developed in which myomas are coagulated rather than removed using electrical energy or laser (thermomyolysis), liquid nitrogen (cryomyolysis), or recently even ultrasound.

Myolysis was performed for the first time by Mergui in France in 1987 using laser YAG to create holes in the myomas resulting in necrosis and narrowing. Later Leukens and Gallinat, in 1993, used bipolar needles from 1 to 3 cm to perform myolysis; their technique was similar to Mergui's.

In 2009 Bettocchi et al. evaluated the efficacy of a procedure to prepare submucosal fibromas with partially intramural development (G1 and G2) >1.5 cm in an outpatient setting (OPPIuM) to facilitate subsequent resectoscope hysteroscopic removal with the patient under general anesthesia.

It has been shown that if the pseudocapsule is removed, the myoma is pushed into the uterine cavity by myometrial contractions. The optimum technique, performed at the time of office hysteroscopy, consisted of incision of the endometrial mucosa and the pseudocapsule covering the myoma, using 5Fr scissors or Versapoint Twizzle bipolar electrode (Gynecare; Ethicon Inc., Somerville, NJ) until the precise identification of the contact surface between the myoma and the pseudocapsule itself. This procedure was intended to facilitate the intramural portion of the myoma protrusion into the cavity during subsequent menstrual cycles and facilitate subsequent resectoscope myomectomy under general anesthesia. Subsequently, in 2013 Haimovich et al. evaluated the feasibility of the same technique using diode laser.

To improve the results obtained in terms of controlled fibroma ablation, the investigators decided to combine the OPPIuM technique and myolysis with a new diode laser: DWLS. The combination of two wavelengths, 980 nm, and 1470 nm, gives a simultaneous absorption in H2O and hemoglobin with excellent hemostasis, cutting, and vaporization capacity, as previously demonstrated in laparoscopic and hysteroscopic surgery.

PURPOSE OF THE STUDY The study aims to examine the feasibility and effectiveness of the OPPIuM technique combined with myolysis using the DWLS diode laser. In addition, to evaluate the reduction of myoma volume and the extent of uterine bleeding with myolysis to improve women's quality of life and avoid resectoscope hysteroscopy for a G2 MIOMA, which may lead to an increase in intraoperative surgical risks and long-term complications.

EXPECTED BENEFITS Compared to the traditional technique (resectoscope hysteroscopic treatment) of G2 myomas, this approach could make the treatment simpler, faster, and in some cases unnecessary.

Compared to the OPPIuM technique with the bipolar electrode and subsequent resectoscope hysteroscopic treatment, the treatment with diode laser could:

1. obtaining the same result and in this case, a subsequent evaluation of comparison between the costs would be useful to evaluate the most suitable instrumentation from a health economics point of view;
2. could obtain a more important clinical result on the patient's symptomatology and volume reduction of myoma, thanks to the well-known properties of tissue vaporization of laser energy, which could avoid the traditional resectoscope hysteroscopic treatment in the operating room burdened with direct health costs and indirect and potential intra-operative or late complications.

INTERVENTION STRATEGY AND INSTRUMENTS The investigators plan to recruit 35 patients who are symptomatic but against hysterectomy and wish to keep the uterus with fibroids ≤ 3 G2. The subjects will be evaluated at the Endometriosis/Pelvic Pain Clinic of the Complex Operating Unit of Gynaecology of the University Hospital of Monserrato and in the other centers involved in the study. All patients will perform a transvaginal examination and ultrasound to provide accurate information on the submucosal myoma characteristics to be operated on and exclude other coexisting uterine or adjunct diseases.

A validated PBAC questionnaire will be filled in to assess the extent of uterine bleeding.

Before carrying out the in vivo test on the enrolled patients, an ex vivo test will be performed on myomas collected during a hysterectomy to evaluate which settings and wave powers are the best to achieve our goal for the myolysis step (the possible decrease in myoma volume).

An office hysteroscopy will be performed in the early proliferative menstrual phase. After a biopsy of the lesion and histological examination, the OPPIuM technique combined with myolysis with the DWLS diode laser using the Myolysis fiber will be performed.

After 1 or 2 menstrual cycles, a transvaginal ultrasound will be performed in the early proliferative phase to assess the volumetric reduction of myoma (following the myolysis). The PBAC questionnaire will be re-administered to assess the clinical response and the extent of uterine bleeding (following the combined technique), and one of the following 3 options will be decided with the patient:

1. do not re-intervene due to a reduction/disappearance of the lesion and/or resolution of the symptomatology
2. perform a second outpatient hysteroscopy to assess the protrusion in the endometrial cavity of the intramural portion of the myoma (following OPPIUM technique) and perform a possible outpatient laser myomectomy
3. program a laser/resettoscopic myomectomy in narcosis. The benefits that the patient can receive derive from the possibility of being able to avoid, thanks to a simple outpatient intervention, the intervention of resectoscope hysteroscopy in narcosis for MIOMA G2, which would lead to increase the intraoperative risks of hemorrhage, cervical trauma, gas embolism, uterine perforation, syndrome from intravasation and late complications such as postoperative intrauterine adhesions and uterine rupture during pregnancy.

The risks associated with the OPPIuM-MYOLYSIS outpatient procedure are, albeit to a very reduced extent compared to resectoscope hysteroscopy, bleeding, and uterine perforation.

With the OPPIuM-MYOLYS technique, complications related to cervical trauma would be avoided (because the cervical canal does not dilate, since the Bettocchi hysteroscope is 4 mm of a much smaller diameter than the resectoscope) and above all, the intravasation syndrome (because of the physiological saline solution at low pressure and for a short time).

Should a narcotic resectoscope hysteroscopy be scheduled due to the first OPPIuM-MYOLYS treatment's failure, the latter will allow surgeons to perform a resectoscope hysteroscopic myomectomy in less than 30 minutes on average, with reduced risks associated with prolonged anesthesia and intravasation syndrome. Furthermore, by favoring the expulsion of MIOMA G2 into the cavity (thus making it G0 or G1), it will be mainly intracavitary lesions, and surgeons will remove these lesions in a single surgical step without intraoperative complications such as uterine perforation, fluid overload, or intraoperative or postoperative bleeding.

POPULATION 35 patients aged between 18 and 48 years with clinical and/or ultrasound diagnosis of uterine fibromatosis, belonging to the Endometriosis/Pelvic Chronic Pain Centre of the Complex Operating Unit of Gynecology of the University Polyclinic of Monserrato and other centers involved in the study. To be eligible for inclusion, patients with ultrasound and hysteroscopic diagnosis of a single submucosal myoma, partially intramural (G1 or G2) ≤ 3 cm, must present symptoms such as abnormal uterine bleeding and pelvic pain, for which surgical treatment was scheduled.

STATISTICAL ANALYSIS The data will be tabulated on a specific database and analyzed using specific software. A descriptive output will be created, and the comparison between variables will be made through parametric and non-parametric tests with a level of significance of 95%. The IBM SPSS Statistics software will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 48 years old
* Diagnosis of symptomatic uterine fibromatosis (abnormal uterine bleeding, pelvic pain and/or infertility) with single fibroma ≤ 3 cm G1 or G2.

Exclusion Criteria:

* Patients who are unable to provide written informed consent or to follow the procedures set out in the protocol.
* Patients with malignant neoplasms or serious systemic diseases
* Patients with multiple fibroids or single > 3 cm
* Asymptomatic patients
* Patients with other uterine or related diseases
* Patients seeking for a pregnancy.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — uterine fibroids
Enrollment: 35 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of symptoms decrease | 3 months
  Change from baseline in symptoms on PBAC score (Herman MC et al.) at 3 months

SECONDARY OUTCOMES:
Evaluation of myoma volume reduction | 3 months
  Change from baseline in moyoma volume on ultrasound at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari,Obstetrics and Gynecological Department,, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stewart EA. Uterine fibroids. Lancet. 2001 Jan 27;357(9252):293-8. doi: 10.1016/S0140-6736(00)03622-9. PMID 11214143
- [Background] Zupi E, Sbracia M, Marconi D, Munro MG. Myolysis of uterine fibroids: is there a role? Clin Obstet Gynecol. 2006 Dec;49(4):821-33. doi: 10.1097/01.grf.0000211961.91616.78. PMID 17082676
- [Background] Bettocchi S, Di Spiezio Sardo A, Ceci O, Nappi L, Guida M, Greco E, Pinto L, Camporiale AL, Nappi C. A new hysteroscopic technique for the preparation of partially intramural myomas in office setting (OPPIuM technique): A pilot study. J Minim Invasive Gynecol. 2009 Nov-Dec;16(6):748-54. doi: 10.1016/j.jmig.2009.07.016. PMID 19896603
- [Background] Haimovich S, Mancebo G, Alameda F, Agramunt S, Sole-Sedeno JM, Hernandez JL, Carreras R. Feasibility of a new two-step procedure for office hysteroscopic resection of submucous myomas: results of a pilot study. Eur J Obstet Gynecol Reprod Biol. 2013 Jun;168(2):191-4. doi: 10.1016/j.ejogrb.2013.01.002. Epub 2013 Jan 31. PMID 23375904
- [Background] Angioni S, Pontis A, Sorrentino F, Nappi L. Bilateral salpingo-oophorectomy and adhesiolysis with single port access laparoscopy and use of diode laser in a BRCA carrier. Eur J Gynaecol Oncol. 2015;36(4):479-81. PMID 26390708
- [Background] Nappi L, Sorrentino F, Angioni S, Pontis A, Litta P, Greco P. Feasibility of hysteroscopic endometrial polypectomy using a new dual wavelengths laser system (DWLS): preliminary results of a pilot study. Arch Gynecol Obstet. 2017 Jan;295(1):3-7. doi: 10.1007/s00404-016-4232-5. Epub 2016 Nov 11. PMID 27834002
- [Background] Herman MC, Mak N, Geomini PM, Winkens B, Mol BW, Bongers MY; International Heavy Menstrual Bleeding IPD Meta-analysis Collaborative Group. Is the Pictorial Blood Loss Assessment Chart (PBAC) score associated with treatment outcome after endometrial ablation for heavy menstrual bleeding? A cohort study. BJOG. 2017 Jan;124(2):277-282. doi: 10.1111/1471-0528.14434. PMID 28012272
- [Background] Di Spiezio Sardo A, Mazzon I, Bramante S, Bettocchi S, Bifulco G, Guida M, Nappi C. Hysteroscopic myomectomy: a comprehensive review of surgical techniques. Hum Reprod Update. 2008 Mar-Apr;14(2):101-19. doi: 10.1093/humupd/dmm041. Epub 2007 Dec 6. PMID 18063608